CLINICAL TRIAL: NCT05779605
Title: Remotely Monitored Rehabilitation in Hemato-oncological Survivors After Treatment: The Tele@Home Study
Brief Title: Telerehabilitation in Hemato-oncological Survivors
Acronym: Tele@home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NU23-09-00048
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy; Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based training (Experimental): 12 weeks of home-based exercise training using modern technology to transfer exercise data remotely. The participants receive a heart rate monitor and sensor. Three sessions per week will be performed (36 sessions overall).
  Interventions: Device: Home-based training
- Center-based training (Active Comparator): 12 weeks of centre-based exercise training under supervision physiotherapists specializing in exercise rehabilitation. The participants receive a heart rate monitor and sensor. The patients in the Center-based training group receive an individually tailored training program on a treadmill and a bicycle ergometer. Three sessions per week will be performed (36 sessions overall).
  Interventions: Device: Center-based training

INTERVENTIONS:
Device: Home-based training — Patients will be instructed to perform three weekly training sessions at home (30 to 50 min/session, at an intensity of 70-85% of their maximum heart rate). Patients in the home training group complete the first three training sessions in the clinic under direct supervision. During these sessions, patients are introduced to the duration and intensity of training. The trainer will provide remote guidance (feedback on training frequency, duration, and intensity) via telephone call once a week. During exercise, patients will use a wearable heart rate monitor (Polar M430, a commercially available device designed for long-term use). Patients will be instructed to properly use the wearable sensor and upload training data to a web-based platform (Polar Flow) via the Internet. Furthermore, patients will be asked to choose their preferred training modality at home (cycling, walking, Nordic walking) and receive instructions and advice.
  Arms: Home-based training
Device: Center-based training — Patients receive three training sessions a week with 30 to 50 min duration at 70 - 90% of their maximal heart rate at the outpatient clinic under direct supervision. Exercise modalities will be walking on a treadmill, riding a bicycle ergometer, and resistance training. Physiotherapists will track the attendance rate and training adherence during the training program.
  Arms: Center-based training

SUMMARY:
This study investigates whether the 12-week home-based exercise training with remote guidance and telemonitoring compared to regular center-based training leads to better long-term cardiorespiratory fitness and physical activity levels in post-treatment patients with lymphoma.

DETAILED DESCRIPTION:
80 lymphoma cancer patients post-treatment (except adjuvant treatment) will be enrolled in the study. Cardiorespiratory fitness (peak oxygen consumption), adverse events, body composition, quality of life, costs and adherence to exercise prescription will be evaluated at baseline, 12-week, and year after enrollment.

Investigators assume that home-based training with remote guidance and telemonitoring with objective training data obtained during rehabilitation after cancer treatment will improve long-term motivation and effectiveness of independent training in cancer survivors, resulting in superior cardiorespiratory fitness and physical activity levels.

ELIGIBILITY:
Inclusion Criteria: Participants

* with hemato-oncological malignancy / lymphoma (in last two months)
* after cancer systemic chemotherapy-based treatment
* with clinically stable state
* with the ability to perform a cardiopulmonary exercise test
* with the ability to understand and write in the Czech language
* with an internet connection at home
* literacy with information and communication technology

Exclusion Criteria: Participants

* with acute heart disease or decompensation in the previous six weeks,
* with psychological severe, cognitive disorders,
* serious training limitations (musculoskeletal disorders)
* currently carried out the recommendations for physical activity (150min per week)
* who take part in a training program under supervision elsewhere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Change from baseline to 12 weeks and 52 weeks
  Peak oxygen uptake during cardiopulmonary exercise test

SECONDARY OUTCOMES:
Health-related quality of life | Change from baseline to 12 weeks and 52 weeks
  Health-related quality of life (SF-36 Form) yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state
Satisfaction - self-completed questionnaire | 12 weeks and 52 weeks
  Subjects will be provided with a 5-item self-completed questionnaire developed by our research team that will measure their satisfaction with the intervention they received and the study in general. The items will be presented in the form of statements to which subjects will be asked to respond using a 1-5 Likert scale ("strongly agree", "agree", "not sure", "disagree", and strongly disagree").
Body water | Change from baseline to 12 weeks and 52 weeks
  Total body water in liters will be measured by bioelectrical impedance analysis.
Muscle mass | Change from baseline to 12 weeks and 52 weeks
  Total muscle mass in kilograms will be measured by bioelectrical impedance analysis.
Body fat percentage | Change from baseline to 12 weeks and 52 weeks
  Body fat percentage will be measured by bioelectrical impedance analysis.
Incidence of exercise adverse events assessed by 5 grade scale | Data will be recorded continuously from the intervention's baseline for 12 weeks and then for 52 weeks
  Participants will be encouraged to use the contact details for reporting incidence of exercise adverse events at any time throughout the study period. The type, incidence, and severity of adverse events by scale (Grade 1: Mild, asymptomatic or mild symptoms; Grade 2: Moderate, minimal; Grade 3: Severe or medically significant; Grade 4: Life-threatening consequences; and Grade 5: Death) will be noted.
Training adherence (Number of compliant participants) | 12 weeks
  Evaluation of the total number of compliant participants (The criterium of compliance with the rehabilitation program is set at 70% of the prescribed training lessons, 100% = 36 lessons)
Maximum Grip Strength | Change from baseline to 12 weeks and 52 weeks
  Maximum grip strength during dynamometer evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ladislav Batalik, Principal Investigator — Department of Rehabilitation, University Hospital Brno, Czech Republic
Locations (1):
- University Hospital Brno, Brno, Czechia

REFERENCES:
- [Derived] Chamradova K, Batalik L, Winnige P, Dosbaba F, Hartman M, Batalikova K, Janikova A, Nehyba S, Felsoci M, Pepera G, Su JJ. Effects of home-based exercise with telehealth guidance in lymphoma cancer survivors entering cardio-oncology rehabilitation: rationale and design of the tele@home study. Cardiooncology. 2024 Jul 30;10(1):46. doi: 10.1186/s40959-024-00249-7. PMID 39080734